CLINICAL TRIAL: NCT06465420
Title: A Phase I Randomized, Observer-blind, Placebo-controlled Trial of a Haemophilus Influenzae Serotype A (Hia) Glycoconjugate Vaccine With Alum Adjuvant in Young Adults 18 to 40 Years of Age
Brief Title: A Study to Evaluate Safety and Immunogenicity of Haemophilus Influenzae Serotype A Vaccine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: InventVacc Biologicals Inc. (Industry)
Collaborators: Hia Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVT 814
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Haemophilus Influenzae Meningitis; Invasive Haemophilus Influenzae Disease
Keywords: Haemophilus influenzae type a meningitis; Indigenous communities; serotype; invasive disease; meningitis; glycoconjugate vaccine; children
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Intervention Model Description: Phase I First-in-Human randomized, controlled study to assess the safety and immunogenicity of the candidate Hia vaccine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the study, the vaccine recipient and those responsible for evaluating any study endpoint (e.g., safety, reactogenicity, and immunogenicity) will all be unaware to which subjects the vaccine was administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine arm (Active Comparator): This arm receives 0.5 mL of a 10 µg dose of Hia Conjugate Vaccine with AdjuPhos.
  Interventions: Biological: Haemophilus influenzae type a (Hia) glycoconjugate vaccine
- Placebo arm (Placebo Comparator): This arm receives 0.5 mL placebo (normal saline).
  Interventions: Biological: Haemophilus influenzae type a (Hia) glycoconjugate vaccine

INTERVENTIONS:
Biological: Haemophilus influenzae type a (Hia) glycoconjugate vaccine — 0.5 mL intramuscular injection, given on days 0 and 28

SUMMARY:
Haemophilus influenzae serotype a (Hia) has emerged as a leading cause of serious illness in Indigenous children in Canada and Alaska in recent decades. In hospital-based surveillance studies, Hia was the most common cause of invasive disease, resulting in morbidity or mortality after Haemophilus influenzae serotype b (Hib). Given the success of the Hib vaccine program and the pathophysiologic similarities between Hib and Hia, immunization is the obvious way to protect Indigenous children living in small and scattered communities. The Public Health Agency of Canada has been working with the National Research Council and other members of the Consortium, including the Canadian Immunization Research Network, McGill Interdisciplinary Initiative in Infection and Immunity, GlycoNet, the Hewitt Foundation, and Inventprise/InventVacc, to develop a Hia vaccine for prevention of this deadly infection. The engagement process initiated by NRC with Consortium members and representatives from Indigenous groups, particularly, has led to the current project plan. In this first-in-human study, the investigators propose investigating the safety and immunogenicity of a novel glycoconjugate candidate vaccine that uses protein carrier CRM197 in healthy adults in the general population. The study will be conducted at the McGill University Health Center Vaccine Study Centre in Montreal and the Canadian Center for Vaccinology in Halifax. The findings of this Phase I study will be necessary to effectively move this potential vaccine solution further along the development continuum.

DETAILED DESCRIPTION:
Haemophilus influenzae serotype a (Hia) can cause invasive diseases, including sepsis and meningitis, similar to serotype b (Hib). In the post-Hib vaccine era, Hia emerged as a prominent cause of invasive infection, largely in Indigenous northern populations in North America. The development of a candidate vaccine to prevent invasive disease due to Hia was initiated by the National Research Council of Canada (NRC) and the Public Health Agency of Canada (PHAC), and the candidate was later licensed to Inventprise/InventVacc Biologicals for further development. Given the success of the Hib vaccine program and the pathophysiologic similarities between Hib and Hia, immunization and the dosing of the Hia vaccine will greatly resemble Hib vaccines. This candidate Hia vaccine will be tested in a randomized, controlled, observer-blind Phase I study in healthy young individuals 18 to 40 years of age from the general population to determine its safety and immunogenicity. This study will be conducted at two sites: the McGill University Health Centre (MUHC) Vaccine Study Centre in Montreal and the Canadian Center for Vaccinology (CCfV) in Halifax; both are study sites of the Canadian Immunization Research Network (Clinical Trials Network). The primary objective of this study is to assess the safety of this novel Hia vaccine. Following vaccine receipt, participants will collect solicited adverse events (AE) in the next 7 days and unsolicited AE for 28 days. Blood for immunogenicity and SBA will be collected on Day 28 after each vaccine dose and on Day 208. Immunogenicity data will be collected as a secondary outcome. The protective capacities of antibodies induced with the Hia vaccine will be directly assessed in vitro with a Hia-specific SBA using a qualified assay developed at the NRC. The SBA titers will be defined as the reciprocal serum dilution required to kill > 50% of the initial bacterial inoculum. Early Hib studies demonstrated the clinical usefulness of a salivary assay for the assessment of mucosal antibody responses during invasive disease and vaccination status once the Hib vaccine was developed. A similar approach can be applied to Hia studies since saliva sampling and testing may provide a non-invasive correlate/surrogate of vaccine-induced immunity that could be very useful in the later-stage development of the vaccine in children and infants. Thus, our Consortium members for Hia have developed a laboratory method for measuring the specific IgA response against Hia-CPS in saliva, which will be used in the exploratory objective. If shown to be safe and immunogenic, and after further consultation and engagement with Indigenous communities, enrolment of Indigenous people in the later phases of the clinical development will be prioritized.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have read, understood, and signed the informed consent form (ICF) prior to participating in the study; the subject must agree to complete study-related procedures and communicate with the study staff at visits and by phone during the study;
2. To be enrolled, subjects must have a body mass index (BMI) ≤ 32 kg/m2 (https://www.cdc.gov/healthyweight/bmi/calculator.html).
3. The subject is considered by the Investigator to be reliable and likely to cooperate with the assessment procedures and be available for the duration of the study;
4. Male and female subjects must be between 18 and 40 years of age at the Vaccination visit (Day 0);
5. Subjects must be in stable health and with no clinically relevant abnormalities that could jeopardize subject safety or interfere with study assessments, as assessed by the Principal Investigator or Sub-Investigator (thereafter referred to as Investigator) and determined by medical history, physical examination, and vital signs; Note: Subjects with a pre-existing chronic disease will be allowed to participate if the disease is stable and, according to the Investigator's judgment, the condition is unlikely to confound the results of the study or pose additional risk to the subject by participating in the study. Stable disease is generally defined as no new onset or exacerbation of pre-existing chronic disease three months prior to vaccination.
6. Female subjects of childbearing potential must have a negative urine pregnancy test result at the Screening and Vaccination visits (Day 0 & 28), and Day 56 and must not be lactating. Non-childbearing females are defined as:

   * Non-ovulating;
   * Surgically-sterile (defined as bilateral tubal ligation, hysterectomy or bilateral oophorectomy performed more than one month prior to vaccination);
   * Post-menopausal (absence of menstruations for 12 consecutive months and age consistent with natural cessation of ovulation);
7. Female subjects of childbearing potential and who are sexually active must use an effective method of contraception for one month prior to vaccination and agree to continue employing adequate birth control measures for at least 60 days post-vaccination. Moreover, female subjects must have no plan to become pregnant for at least two months post-vaccination. Abstinent subjects who are ovulating should be asked what method(s) they would use should their circumstances change, and subjects without a well-defined plan should be excluded. The following relationship or methods of contraception are considered to be effective:

   * Hormonal contraceptives (e.g., oral, injectable, topical [patch], or estrogenic vaginal ring);
   * Intra-uterine device with or without hormonal release;
   * Male partner using a condom plus spermicide or sterilized partner (at least one year prior to vaccination);
   * Credible self-reported history of heterosexual vaginal intercourse abstinence until at least 60 days post-vaccination;
   * Female partner.
8. The overall similarity of the Hia candidate vaccine to Hib vaccines widely administered in multiple doses to infants for several decades and the absence of genotoxicity in the toxicity study provides further reassurance that a contraceptive requirement in males is not needed.

Exclusion Criteria:

1. According to the Investigator's opinion, history of an ongoing acute or evolving medical or neuropsychiatric illness. "Evolving" is defined as:

   * Requiring a new medical or surgical treatment during the three months prior to study vaccine administration unless the criteria outlined in inclusion criterion no. 5 can be met (i.e., the Investigator can justify inclusion based upon the innocuous nature of medical/surgical events and/or treatments);
   * Requiring any significant change in a chronic medication (i.e., drug, dose, frequency) during the three months prior to study vaccine administration due to uncontrolled symptoms or drug toxicity unless the innocuous nature of the medication change meets the criteria outlined in inclusion criterion no. 5 and is appropriately justified in writing by the Investigator in the source document.
2. Any medical or neuropsychiatric condition or any history of excessive alcohol use or drug abuse that would render the subject unable to provide informed consent or unable to provide valid safety observations and reporting, including methadone (methadone as treatment for opioid dependence may be acceptable if the subject has been otherwise opioid-free for at least three years);
3. A history of neurologic disorders or seizures;
4. Any history of autoimmune disease other than hypothyroidism on stable replacement therapy (including, but not limited to rheumatoid arthritis, systemic lupus erythematosus, Crohn's disease, type 1 diabetes, and inflammatory bowel disease) or any confirmed or suspected congenital or acquired immunosuppressive condition or immunodeficiency including known or suspected human immunodeficiency virus (HIV), hepatitis B or C infection, the presence of lymphoproliferative disease, tested for at the screening. Very little investigator discretion will be permitted with this exclusion criterion but rare subjects may still be eligible to participate with appropriate written justification in the source document (e.g., documented HBV carrier status with no evidence of active liver disease, cured HCV with documented clearance of virus, very mild psoriasis [i.e., a small number of minor plaques requiring no treatment], etc.);
5. Any hematologic or biochemical laboratory abnormalities, as defined by lab normal ranges. To exclude transient abnormalities, the Investigator may repeat a test once, and if the repeat test is normal according to local reference ranges, participant may be enrolled. Grade 1 abnormalities of laboratory values will not be exclusionary if considered not clinically significant by the Investigator.
6. Any history of status asthmaticus or ongoing serious problems with asthma, hospitalization for asthma control, or recurrent asthma episodes requiring medical attention in the last three years (one or more episodes per year);
7. Administration or planned administration of any vaccine (including routine vaccines) within 30 days prior to Hia immunization and up to 30 days post-second dose of vaccine. Immunization on an emergency basis will be evaluated case-by-case by the Investigator;
8. Administration of any adjuvanted, "standard" influenza non-adjuvanted (e.g., live attenuated inactivated vaccine or split inactivated vaccine administered by intranasal, intradermal, or intramuscular [IM] route) or investigational vaccine within 30 days prior to randomization, administration prior to the completion of the study and up to 30 days post-second dose of vaccine;
9. Use of any investigational or non-registered product within 30 days or five half-lives, whichever is longer, prior to randomization or planned use during the study period. Subjects may not participate in any other investigational or marketed drug study while participating in this study;
10. Treatment with systemic glucocorticoids at a dose exceeding 10 mg of prednisone (or equivalent) per day for more than seven consecutive days or for ten or more days in total, within one month of study vaccine administration; any other cytotoxic or immunosuppressant drug, or any immunoglobulin preparation within three months of vaccination and until the completion of the study. Low doses of nasal or inhaled glucocorticoids are allowed. Topical steroids are permitted;
11. Any significant disorder of coagulation including, but not limited to, treatment with warfarin derivatives or heparin. Persons receiving prophylactic anti-platelet medications (e.g., low-dose aspirin [no more than 81 mg/day]), and without a clinically apparent bleeding tendency are eligible. Subjects treated with new generation drugs that do not increase the risk of IM bleeding (e.g., clopidogrel) are also eligible;
12. History of allergy to any of the constituents of the Hia Conjugate Vaccine or a history of anaphylaxis to any vaccines;
13. History of anaphylactic allergic reactions to Hia Conjugate Vaccine components;
14. Use of antihistamines within 48 hours prior to study vaccination;
15. Use of prophylactic medications (e.g., acetaminophen/paracetamol, aspirin, naproxen, or ibuprofen) within 24 hours of randomization to prevent or pre-empt symptoms due to vaccination or if they are on recurring doses of these medications for other reasons;
16. Have a rash, dermatological condition, tattoos (a tattoo on one deltoid only is acceptable), muscle mass, or any other abnormalities at the injection site that may interfere with injection site reaction rating;
17. Subjects who have received blood-derived products or a blood transfusion within 90 days prior to study vaccination;
18. Subjects with abnormal age-specific vital signs. For adults >18 years of age: systolic blood pressure [BP] ≥ 140 mmHg and/or diastolic [BP] ≥ 90 mmHg; heart rate [HR] ≤ 45 beats/min and ≥ 100 beats/min evaluated by an Investigator to be clinically significant. A subject with abnormal vital signs results may be included in the study based on Investigator's judgment (e.g., a resting [HR] ≤ 45 in highly trained athletes).
19. Presence of any febrile illness (including an oral temperature [OT] ≥ 38.0 ˚C within 24 hours prior to vaccination);
20. Cancer or treatment for cancer within three years prior to study vaccine administration. Persons with a history of cancer who are disease-free without treatment for three years or more are eligible. However, individuals with conditions such as treated and uncomplicated basal cell carcinoma of the skin or non-treated, non-disseminated local prostate cancer may be eligible;
21. Subjects identified as an Investigator or employee of the Investigator or clinical site with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse) of the Investigator or any employee of InventVacc (or their family members);
22. Subjects with a history of Guillain-Barré Syndrome.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Percentage, intensity, and relationship of adverse events to vaccination | Solicited AEs for 7 days and unsolicited AEs for 28 days after each of two IM doses 28 days apart; SAEs and MAAEs up to 6 months
  Solicited adverse events (AEs) and unsolicited AEs, serious adverse events (SAEs) and medically attended adverse events (MAAEs)

SECONDARY OUTCOMES:
Immunogenicity | Measure the levels of anti-Hia capsular polysaccharide 28 days after each of two doses and at 180 days post-second dose (Days 0, 28, 56, and 208).
  Anti-Hia CPS-specific IgG and serum bactericidal assay (SBA)

OTHER OUTCOMES:
Immunogenicity | 28 days after each of two doses and at 180 days post-second dose (Days 0, 28, 56, and 208)
  Measure anti-Hia CPS specific IgA by ELISA in the saliva

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ward, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Joanne Langley, MD, Principal Investigator — Canadian Center for Vaccinology; Scott Halperin, MD, Principal Investigator — Canadian Center for Vaccinology
Locations (2):
- Canada (2):
  - Canadian Center for Vaccinology (CCfV), Halifax, Nova Scotia
  - McGill University Health Centre (MUHC) Vaccine Study Centre, Montreal, Quebec